CLINICAL TRIAL: NCT06337084
Title: Open Label Pilot Study Evaluating Diagnostic Efficacy and Dosimetry of MNPR-101-DFO*-89Zr in Patients With Solid Tumors
Brief Title: Diagnostic Efficacy and Dosimetry of MNPR-101-DFO*-89Zr in Patients With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Monopar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: MNPR-101-D001
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Solid Tumor, Adult; Bladder Cancer; Urothelial Carcinoma; Triple-negative Breast Cancer; Lung Cancer; Colorectal Cancer; Gastric Cancer; Ovarian Cancer; Pancreatic Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell; Triple Negative Breast Neoplasms; Lung Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- MNPR-101-DFO*-89Zr Single Infusion and PET/CT Imaging (Experimental): Participants receive a single injection of MNPR-101-DFO*-89Zr on Day 1 with administered activity between 37-74 MBq (or 1-2 mCi). PET/CT imaging will occur post-infusion at 2 h (Day 1), once on Days 3-5, and once on Days 7-10.
  Interventions: Drug: MNPR-101-DFO*-89Zr; Diagnostic Test: PET/CT Diagnostic Imaging

INTERVENTIONS:
Drug: MNPR-101-DFO*-89Zr — Participants will receive one dose of MNPR-101-DFO*-89Zr infused intravenously on Day 1 for PET scans
Diagnostic Test: PET/CT Diagnostic Imaging — PET/CT imaging will occur post-infusion at 2 h (Day 1), once on Days 3-5, and once on Days 7-10 for tumor lesion observation.

SUMMARY:
This is an open-label pilot study of a new PET/CT imaging agent MNPR-101-DFO*-89Zr in patients with solid tumor cancers. These cancers may include bladder/urothelial, triple-negative breast, lung, colorectal, gastric, ovarian, and pancreatic cancers.

MNPR-101-DFO*-89Zr is made of MNPR-101, a humanized IgG1 monoclonal antibody and a radioisotope Zirconium-89. This imaging agent may show where tumors are present in the body using a PET-scan.

Participants will be injected with the radioactive tracer once. After injection, participants will have 3 PET-scans. Each PET-scan will take about 30 minutes. The PET-scans are on separate days within 10 days after injection (e.g., 2 hours after injection, plus 3-5 days and 7-10 days after injection). Furthermore, the investigators will take blood samples 6 times (5 mL each). Blood pharmacokinetics (PK) will be measured on Day 1 at 10 min, 1h, 2h, once on Days 3-5, and once on Days 7-10.

The study will see if the new imaging agent correctly shows all tumors. In the future, this method may be useful to help predict who will benefit from certain therapies.

DETAILED DESCRIPTION:
This is an open-label, multi-center, imaging, and dosimetry pilot study to evaluate MNPR-101-DFO*-89Zr, a radiolabeled tracer composed of humanized IgG1 monoclonal antibody MNPR-101 which targets cancers that express the urokinase plasminogen activator receptor (uPAR) used with Positron Emission Tomography/Computed Tomography (PET/CT) imaging in patients with solid tumor cancers.

The study aims to determine the dosimetry and biodistribution, tumor standard uptake values (SUV), safety profile, and blood pharmacokinetics (PK) of MNPR-101-DFO*-89Zr.

On Day 1, patients will receive a single infusion of MNPR-101-DFO*-89Zr. All subjects will receive 37 to 74 MBq (1-2 mCi) of 89Zr with radioactivity determined based upon the site's PET/CT equipment. The antibody mass dose of MNPR-101-DFO*-89Zr will be increased in a stepwise fashion to a maximum of 80 mg. Before increasing to the next mass antibody dose level, each cohort of 2 patients will be assessed following the Day 7-10 visit for related hematologic or hepatologic events reported as CTCAE Grade 4, or CTCAE Grade 3 if lasting longer than 30 days.

PET/CT imaging will occur post-infusion at 2 h (Day 1), once on Days 3-5, and once on Days 7-10. PK blood sampling, for analysis via well or gamma counter, will occur post-infusion on Day 1 at 10 min, 1h, 2h, once on Days 3-5, and once on Days 7-10.

Dosimetry will be calculated using OLINDA/EXM or a similar software. Tumor SUVs will be assessed and compared to a prior 18F-FDG PET scan. PK measurements will be made via well or gamma counter and adjusted for radioactive decay.

The primary endpoints will assess dosimetry, biodistribution including target safety organs (e.g., liver, kidney, bone marrow, and lungs), tumor SUV, and the safety profile of MNPR-101-DFO*-89Zr. Patients will be followed for 1-month post infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and/or cytologically confirmed solid tumor cancer.
2. Age ≥18 years.
3. Measurable disease ≥ 1 cm on prior 18F-FDG PET/CT scan. Up to 4 subjects may be enrolled with FDG-avid disease which do not meet ≥ 1 cm measurement on CT.
4. Ability to understand and willingness to sign a written informed consent document.
5. A prior standard-of-care 18F-FDG PET/CT scan within past 60 days.
6. Tumor sample available for IHC testing to demonstrate uPAR expression.
7. Females of childbearing potential must have a negative serum pregnancy test at time of screening and a negative urine pregnancy test on Day 1 prior to study drug administration if screening is >7 days prior to Day 1. A rapid serum pregnancy test result performed as standard-of-care will be accepted if available.
8. Both males and females must agree to use highly effective contraceptive precautions if conception is possible during the dosing period and up to 1 month after dosing.
9. Female patients who are lactating must agree to discontinue breastfeeding prior to the dose of study drug and must refrain from breastfeeding for 1 month following the last dose of study drug.

Exclusion Criteria:

1. Chemotherapy, radiotherapy (other than short cycle of palliative radiotherapy), or immunotherapy within 14 days prior to administration of MNPR-101-DFO*-89Zr, or continuing adverse effects (>grade 1, excluding alopecia, anorexia, fatigue, and neuropathy) from such therapy (Common Terminology Criteria for Adverse Events [CTCAE] version 5.0).
2. Prior treatment with any radiopharmaceutical or investigational agents within 4 weeks or 5 effective half-lives, whichever is longer, prior to administration of the first dose of MNPR-101-DFO*-89Zr.
3. Have evidence of impaired organ function at Screening and within 1 week prior to dosing MNPR-101-DFO*-89Zr, particularly:

   * Bone marrow i. Platelets <75 K/mcL. ii. ANC <1.0 K/mcL.
   * Liver function i. AST/ALT >2.5xULN (institutional upper limits of normal) OR >5×ULN for patients with liver metastases.

   ii. Bilirubin >1.5xULN OR >3×ULN for patients with known Gilbert's Syndrome.
   * Renal function i. eGFR ≤45 mL/min determined using BSA-adjusted Chronic Kidney Disease Epidemiology Collaboration CKD-EPI 2021 formula [https://www.kidney.org/professionals/kdoqi/gfr_calculator].
4. Other serious, non-malignant diseases that may interfere (e.g., renal, hepatic, or hematologic) with the objectives of the study, safety, or compliance, as judged by the investigator.
5. Cognitive impairment or contraindications that may compromise the ability to give informed consent or comply with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
To assess dosimetry and biodistribution of MNPR-101-DFO*-89Zr | Post infusion at 2 h on Day 1, once on Days 3-5, and once on Days 7-10.
  The biodistribution of MNPR-101-DFO*-89Zr is assessed via PET/CT imaging scans, particularly of target safety organs (e.g., liver, kidney, red marrow, and lungs). Dosimetry is calculated using OLINDA/EXM or a similar software.
To assess tumor Standard Uptake Value (SUV) of MNPR-101-DFO*-89Zr | Post infusion at 2 h on Day 1, once on Days 3-5, and once on Days 7-10.
  Tumor SUV is measured via PET/CT imaging by calculating the amount of radiotracer uptake in identified tumors. SUV mean, max, and peak of the tumors will be summarized at each timepoint per subject. Tumor SUV will be analyzed between subjects with the same cancer type as well as between cancer types.
To assess safety of MNPR-101-DFO*-89Zr as assessed by CTCAE 5.0 | Screening through Day 30 Safety Visit.
  The safety profile of MNPR-101-DFO*-89Zr will be determined through assessment of adverse event (AE) type, incidence, severity, time of appearance, and related causes (detected by physical explorations and laboratory tests). Adverse events will be graded and tabulated using NCI CTCAE v5.0.

SECONDARY OUTCOMES:
To assess pharmacokinetics (PK) of MNPR-101-DFO*-89Zr via well or gamma counter | Post infusion at 10 min, 1 h and 2 h on Day 1, once on Days 3-5, and once on Days 7-10.
  PK, mean and standard deviation plasma drug concentration are collected and measured via well or gamma counter to assess the imaging agent's interaction in blood and/or serum at each timepoint per subject.

OTHER OUTCOMES:
To assess tumor uptake to background and tumor uptake to liver ratios | Post infusion at 2 h on Day 1, once on Days 3-5, and once on Days 7-10.
  Tumor to background (skeletal muscle) and tumor to liver uptake ratios using PET/CT imaging will be calculated from the lesion-free volume of interest (VOI) (reference tissue) using SUV_mean_lesion / SUV_mean_reference.
To assess benefit of added cold MNPR-101 antibody | Post infusion at 10 min, 1 h and 2 h on Day 1, once on Days 3-5, and once on Days 7-10.
  Determination of optimal cold antibody will be assessed based on the level of cold antibody where PK values in blood plateau and behave approximately linearly on a log scale over time, using time-corrected gamma counts of whole blood and/or serum.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Rod Hicks, MD, Principal Investigator — Melbourne Theranostic Innovation Centre (MTIC)
Locations (1):
- Melbourne Theranostic Innovation Centre (MTIC), North Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No